CLINICAL TRIAL: NCT05823142
Title: Health Behavior Intervention for Adults With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Stephanie Griggs, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025P011836; R01DK136604 (NIH); STUDY20230448 (Other: Case Western)
Record Dates: First submitted 2023-04-04; First posted 2023-04-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Intervention Model Description: Behavioral: Sleep Self-Management
Who Masked: Participant
Masking Description: Both conditions will receive time-balanced sessions with the study team. Participants will not be told whether in the experimental condition or the condition delivering usual care until after the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CB-sleep (Experimental): Initial instruction for the CB-sleep intervention will occur 60-minute telehealth session. The initial action planning session with a sleep report and booster sessions will be interactive and stage matched. The intervention will include an interactive PowerPoint with the participant's clinician sleep report with personalized feedback. They will be encouraged to systematically extend their time in bed by 1 hour and maintain the extension on both weekends and weekdays. Weekly titration will occur according to the following parameters: if sleep efficiency is ≥ 85%, time in bed is increased by 15 minutes per week until a total of a 1 hour increase in time in bed is achieved, if sleep efficiency is <85%, time in bed remains the same. There will be weekly follow-ups (email, phone, text, video chat) and telehealth 4-week booster sessions. Sleep reports generated by the baseline actigraphy report will be shared with participants with brief action planning and goal setting.
  Interventions: Behavioral: CB Sleep
- Attention Control Enhanced Usual Care arm (No Intervention): After baseline, the RA assigned to this condition will schedule a 60-minute telehealth appointment to provide instruction for enhanced usual care at the initial consultation visit via contact at T1 (60-minute telehealth session in a private location). The time-balanced follow-up sessions will remain neutral and focused on health perceptions, current plan of care, and relationship building as opposed to the CB-sleep condition's focus on sleep promotion and extension. The RA assigned to the control condition will ask participants to (a) describe how they are doing and (b) ask how confident they are in achieving the goals they have set for themselves. These calls will help to build a relationship with participants to promote study retention. The investigators recognize that participants may obtain self-initiated diabetes self-management in this group, which will vary and will use a Diabetes Self-Management Tracking Form to monitor weekly information acquisition.

INTERVENTIONS:
Behavioral: CB Sleep — The CB-sleep intervention is a cognitive behavioral intervention guided by principles and practices from motivational interviewing and the psychology of behavior change, primarily drawing on self-efficacy and action planning theory. The goals of CB-sleep are for participants to achieve adequate sleep duration (7-9 hours per night), adequate sleep efficiency (≥ 85%), and regular sleep timing (<60-minute differences in bed and wake times). The intervention components include improving sleep knowledge (hygiene), developing a nightly routine, addressing competing activities, modifying environmental conditions, lifestyle (avoiding caffeine and vigorous exercise before bed), technology (limiting or avoiding screens for at least one hour before bed), basic stress-management (progressive muscle relaxation and guided imagery), and self- monitoring.
  Arms: CB-sleep

SUMMARY:
Type 1 diabetes (T1D) affects approximately 2 million Americans, and only 2 in 8 young adults ages 18-31 years achieve glycemic targets (glycated hemoglobin A1C <7.0%). Achieving glycemic targets is associated with reduced risk of micro-and macrovascular complications. Sleep deprivation leads to impaired glucose tolerance and insulin sensitivity in adults without chronic conditions and with T1D. Promoting sleep in laboratory and natural environments contributes to improvements in insulin sensitivity, glucose levels, and distress symptoms in young adults without chronic conditions and more time in range in adolescents with T1D. Multiple dimensions of sleep health (alertness, timing, efficiency, and sleep duration) are associated with better achievement of glycemic targets in adults with T1D. Therefore, sleep health dimensions are appropriate therapeutic targets to improve glucoregulation and other diabetes self-management outcomes in this population.

Our primary objective is to evaluate the immediate and short-term effects of a 12-week CB-sleep intervention compared to enhanced usual care (time balanced attention control) on actigraphy- and self-report derived sleep health dimensions and diabetes self-management outcomes (glycemia and distress symptoms) over 9-months (Stage II of the NIH Model for Behavior Change, ORBIT phase III). CB-sleep is guided by principles and practices from motivational interviewing and the Transtheoretical Model of Behavior Change with interactive stage-matched sessions.

DETAILED DESCRIPTION:
Overview: The investigators will conduct a powered randomized controlled trial (RCT) and recruit a contemporary cohort of 248 young adults with T1D and randomly assign them to one of two conditions: CB-sleep or a time-balanced attention control (enhanced usual care) condition. The study will evaluate the immediate and short-term effects of CB-sleep compared to enhanced usual care on actigraphy and self-report derived sleep health dimensions (aim 1), glycemia and other diabetes self-management outcomes (aim 2), and whether sleep health mediates associations between the CB-sleep and enhanced usual care conditions (aim 3). All participants will complete a battery of validated questionnaires and objective measures of sleep and glycemia captured at baseline to post-intervention (3 months) and at a 6- and 9-month follow-up.

Study Design:

A two-arm, RCT will be used to evaluate the efficacy of CB-sleep compared to a time-balanced attention control condition (enhanced usual care). Data collection will include T0 baseline measures (questionnaires and 14-days of sleep/glucose monitoring), T1 will include the allocation to the experimental or control condition, T2 will include immediate post baseline measures at 3-months, T3 will include repeating measures at 6-months, and T4 will include repeating measures at 9-months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 40 years
* Type 1 Diabetes at least 1 year
* One or more sleep health dimension out of range

Exclusion Criteria:

* Non-English speaking
* A1C < 7% or >80% time in glucose range

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Multidimensional sleep health composite score | Baseline, 3, 6 and 9 months post-intervention
  The multidimensional sleep health composite score will measure sleep regularity, satisfaction, alertness, timing, efficiency, and duration of sleep. The total possible score range is 0-6 with higher scores indicating higher or better sleep health.
Glycated hemoglobin (HbA1C) | Baseline, 3, 6 and 9 months post-intervention
  Changes in glycemia will be measured by glycated hemoglobin (HbA1C) at baseline, 3, 6 and 9 months.

SECONDARY OUTCOMES:
Glucose variability | Baseline, 3, 6 and 9 months post-intervention
  % coefficient of variation will be measured by Continuous glucose monitor (CGM) or glucose meter
Time in range (70-140 mg/dL) | Baseline, 3, 6 and 9 months post-intervention
  Time in rage for glycemic control (70-140 mg/dL) will be measured by Continuous glucose monitor (CGM) or glucose meter
General distress symptoms | Baseline, 3, 6 and 9 months post-intervention
  PROMIS v1.0 Emotional Distress (Cronbach's α = 0.95, ICC 0.69 to 0.88), With a standardized normative T-score of 50 and a standard deviation of 10, T-scores <55 would translate as normal; 55-60 as mild; 60-70 as moderate, and ≥70 as severe distress
Diabetes distress symptoms | Baseline, 3, 6 and 9 months post-intervention
  Diabetes Distress Scale (Cronbach's α = 0.88 to 0.93, ICC 0.44 to 0.64), Average score of < 2.0 = reflects little or no distress Average score between 2.0 and 2.9 = reflects moderate distress, Average score > 3.0 = reflects high distress, A total or subscale score > 2.0 (moderate distress) is considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Griggs, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No